CLINICAL TRIAL: NCT06422442
Title: Information Processing Biases in Adults Who Stutter: Behavioral and Eye-tracking Indices of Threat-related Attention Allocation
Brief Title: Information Processing Biases in Adults Who Stutter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R21DC020557 (NIH)
Record Dates: First submitted 2024-05-13; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Stuttering, Adult
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Masking Description: Individuals reviewing and coding data will not be aware of group status or diagnoses for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye tracking tasks (Experimental): All participants complete three tasks in which they view threat-related and neutral stimuli (words or faces)
  Interventions: Behavioral: Threat-related stimulus exposure

INTERVENTIONS:
Behavioral: Threat-related stimulus exposure — Participants will view threat-related stimuli (words or faces) paired with nonthreat matches in three related experimental paradigms.

SUMMARY:
The goal of this clinical trial is to examine whether stuttering is associated with a tendency to attend more quickly or for longer durations to threat-related information in the environment (threat-related attention bias). The main questions it aims to answer are:

Do adults who stutter, relative to adults who do not stutter, attend to threat-related stimuli more than neutral information? Are attentional biases observed across different types of threat or are they specific to threats related to stuttering experiences? Do measures of attention bias explain individual differences in psychological reactions among adults who stutter?

DETAILED DESCRIPTION:
The goal of the project is to examine threat-related attentional processes associated with stuttering. In Aim 1, investigators will establish differences in attention bias (AB) in adults who do and do not stutter and the processing stage at which differences emerge. In Aim 2, investigators will compare AB effects across different categories of threat stimuli to determine whether threat-related AB in adults who stutter is general or disorder-specific. In Aim 3, the investigators examine the role of AB as a causal factor mediating effects of individual risk-factors (related to temperament and attention control) on stuttering impact and anticipation. Participants will include 35 adults who stutter and 35 adults who stutter between the ages of 18-30 years, all meeting specified eligibility criteria. All participants will complete three experimental tasks for measuring AB: (1) a free-viewing task, (2) dot-probe task, and (3) emotional Stroop task. Study procedures will be administered over two sessions (2-2.5 hours each) scheduled within three weeks of each other. Key outcomes will include reaction time and eye-tracking measures, which will be used to extract multiple AB indices. Data will be analyzed via mixed-effects regression analysis with a random intercept for subject and maximal converging random-slopes structure. Age, gender, socioeconomic status and various measures used for inclusion purposes will be included as covariates. Mediation analyses will assess four relationships (Temperament -> Stuttering impact, Temperament -> Anticipation, Attention control -> Stuttering impact, and Attention control -> Anticipation), with AB as the mediator variable in each analysis.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English as their primary language
* Normal hearing (based on pure tone screening)
* Normal or corrected vision (based on report)
* Normal color vision (based on Ishihara Test, Concise Edition)
* Nonverbal intelligence within at least average range based on Test of Nonverbal Intelligence, 4th Edition
* Expressive language within at least average range score based on Expressive One-Word Picture Vocabulary Test

Additional inclusion criteria for adults who stutter:

* Self-identification as a person who stutters
* Score of at least 11 (mild stuttering) on Stuttering Severity Index, 4th Edition

Exclusion Criteria:

* Reported significant medical history
* Psychological or emotional disorder
* History of frank neurological injury
* Known speech, language, or learning disorder(s) other than stuttering
* Reading difficulties
* Score within clinically significant range for ADHD on Adults ADHD Self-Rating Scale
* Score within clinically significant range for depression on Beck Depression Inventory
* Score within clinically significant range for anxiety on State-Trait Anxiety Inventory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reaction time (RT) measures | Trial duration (maximum of 10 seconds)
  A) A key outcome measure from the dot-probe task will consist of RTs for congruent trials (in which probe appears in the location of threat stimulus) vs. incongruent trials (probe replaces neutral stimulus). (B) Key outcome measure from the emotional Stroop will include RT for threat vs. neutral words.
Total dwell time on threat | Trial duration (8 seconds)
  This primary (and most reliable) index of AB will be extracted from eye movement data and represents the total duration of all fixations to areas of interest with threat stimuli for each trial of the free-viewing task.

SECONDARY OUTCOMES:
Eye tracking indices of AB | Trial duration (8 seconds)
  Additional indices of AB will be extracted from eye movement data and examined in exploratory manner: (1) probability of first fixation to an area of of interest (AOI), (2) first fixation latency, (3) first fixation duration, 4) first-run dwell time (representing summed duration of all fixations to an AOI from the first fixation until the AOI is exited), and (5) second-run dwell time (summed duration of all fixations within an AOI from the second time the AOI is entered until it is exited).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made freely and publicly available on OSF (https://osf.io) together with our publications, with prior Institutional Review Board approval. Archived data will also be made available to other researchers upon request (by emailing the PI) and without cost. A signed data-sharing agreement will be required for researchers to access data; the agreement will stipulate that shared data must be used solely for the purpose of research, must not be transferred to or shared with others, must not be manipulated for the purpose of identifying subjects, and that the planned research must be reviewed and approved by an Institutional Review Board.